CLINICAL TRIAL: NCT02354586
Title: A Phase 2, Open-Label, Single-Arm Study to Evaluate the Safety and Efficacy of Niraparib in Patients With Advanced, Relapsed, High-Grade Serous Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer Who Have Received Three or Four Previous Chemotherapy Regimens
Brief Title: A Study of Niraparib in Patients With Ovarian Cancer Who Have Received Three or Four Previous Chemotherapy Regimens
Acronym: QUADRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tesaro, Inc. (Industry)
Collaborators: Facing Our Risk of Cancer Empowered (Other); Myriad Genetics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 213360; PR-30-5020-C (Other: Tesaro)
Record Dates: First submitted 2015-01-23; First posted 2015-02-03 (Estimated); Results first posted 2020-04-09 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-07

CONDITIONS: Ovarian Neoplasms; Ovarian Cancer
Keywords: gBRCAmut; BRCA; PARP inhibitor; HRD; Ovarian cancer; Serous Epithelial; Fallopian Tube; Primary Peritoneal
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib

ARMS (1):
- Niraparib (Experimental)
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib

SUMMARY:
This is a Phase 2, open-label, single arm study to evaluate the safety and efficacy of niraparib in ovarian cancer patients who have received three or four previous chemotherapy regimens. Niraparib is an orally active PARP inhibitor. Niraparib will be administered once daily continuously during a 28-day cycle. Health-related quality of life will be measured by Eastern Cooperative Oncology Group performance status (ECOG). Safety and tolerability will be assessed by clinical review of adverse events (AEs), physical examinations, electrocardiograms (ECGs), RECIST tumor assessments and safety laboratory values.

ELIGIBILITY:
Inclusion Criteria:

* Patients must agree to undergo tumor HRD testing and blood gBRCAmut status testing.
* Patients of childbearing potential must have negative pregnancy serum test within 72 hours of being dosed
* Patients must have histologically diagnosed high-grade (Grade 2 or 3) serous epithelial ovarian, fallopian tube, or primary peritoneal cancer with recurrent disease and must have been previously treated with chemotherapy and experienced a response lasting at least 6 months to first-line platinum based therapy.
* Patients Must have completed 3 or 4 previous chemotherapy regimens.
* Patients must have completed their last chemotherapy regimen > 4 weeks prior to treatment initiation.
* Patients must have measurable disease according to RECIST (v.1.1).
* Patients must have formalin-fixed, paraffin-embedded tumor samples available from the primary or recurrent cancer or agree to undergo fresh biopsy prior to study treatment initiation.
* Patients must agree to blood samples during screening and at the end of treatment for cytogenetic analysis.

Exclusion Criteria:

* Patients must not have any known, persistent (> 4 weeks), ≥Grade 3 hematologic toxicity during the last cancer therapy. Patients must not have any known, persistent (>4 weeks), ≥ Grade 3 fatigue during the last cancer therapy.
* Patients must not have received pelvic radiotherapy as treatment for primary or recurrent disease within 1 year of the first dose of study treatment.
* Patients must not have symptomatic uncontrolled brain or leptomeningeal metastases.
* Patients must not be considered a poor medical risk due to a serious, uncontrolled medical disorder, nonmalignant systemic disease or active, uncontrolled infection.
* Patients must not have received a transfusion (platelets or red blood cells) within 4 weeks of the first dose of study treatment.
* Patients must not have known history or current diagnosis of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2015-03-23 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2021-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (48):
- United States (44):
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Burbank, California
  - GSK Investigational Site, Duarte, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Santa Barbara, California
  - GSK Investigational Site, Stanford, California
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Covington, Louisiana
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Burlington, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, Hackensack, New Jersey
  - GSK Investigational Site, Morristown, New Jersey
  - GSK Investigational Site, East Setauket, New York
  - GSK Investigational Site, Jamaica, New York
  - GSK Investigational Site, Lake Success, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Wynnewood, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, The Woodlands, Texas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Tacoma, Washington
- Canada (4):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec

REFERENCES:
- [Background] Moore KN, Secord AA, Geller MA, Miller DS, Cloven N, Fleming GF, Wahner Hendrickson AE, Azodi M, DiSilvestro P, Oza AM, Cristea M, Berek JS, Chan JK, Rimel BJ, Matei DE, Li Y, Sun K, Luptakova K, Matulonis UA, Monk BJ. Niraparib monotherapy for late-line treatment of ovarian cancer (QUADRA): a multicentre, open-label, single-arm, phase 2 trial. Lancet Oncol. 2019 May;20(5):636-648. doi: 10.1016/S1470-2045(19)30029-4. Epub 2019 Apr 1. PMID 30948273
- [Derived] Monk BJ, Romero I, Graybill W, Churruca C, O'Malley DM, Knudsen AO, Yap OWS, Baurain JF, Rose PG, Denys H, Ghamande S, Pisano C, Fabbro M, Braicu EI, Calvert PM, Amit A, Prendergast E, Taylor A, Kheibarshekan L, Zhang ZY, Zajic S, Jewell RC, Gupta D, Gonzalez-Martin A. Niraparib Population Pharmacokinetics and Exposure-Response Relationships in Patients With Newly Diagnosed Advanced Ovarian Cancer. Clin Ther. 2024 Aug;46(8):612-621. doi: 10.1016/j.clinthera.2024.06.001. Epub 2024 Jul 16. PMID 39019698

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, single arm study to evaluate the safety and efficacy of niraparib in ovarian cancer participants who have received previous chemotherapy regimens.
Pre-assignment Details: A total of 463 participants were enrolled in the study (Safety Population was comprised of all participants who received at least 1 dose of study drug).
Groups:
- Niraparib 300 mg: Participants received Niraparib (300 milligram [mg], taken as 3 capsules of 100 mg once daily [QD]) orally beginning on Day 1 of every cycle (28 days) until treatment discontinuation.
Period: Overall Study
Arm/Group | Niraparib 300 mg
Started | 463
Completed | 0
Not Completed | 463
Not completed — Death | 230
Not completed — Withdrawal by Subject | 59
Not completed — Lost to Follow-up | 11
Not completed — Sponsor decision | 51
Not completed — Site closure | 2
Not completed — Intercurrent illness | 1
Not completed — Protocol Violation | 3
Not completed — Physician Decision | 13
Not completed — Lack of Efficacy | 86
Not completed — Adverse Event | 7

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were reported for Safety Population.
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 463
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.3 (9.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 463
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 394
  Black | 20
  Asian | 16
  American Indian or Alaska Native | 1
  Unknown | 32

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: The ORR was defined as the percentage of participants achieving complete response (CR) or partial response (PR) as assessed by the Investigator per Response Evaluation Criteria in Solid Tumors (RECIST) (version1.1), where CR=Disappearance of all target lesions. Any pathological lymph nodes must be <10 millimeters (mm) in the short axis, PR=At least a 30 percent (%) decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters. Primary Analysis Population comprised of participants who received 3 or 4 prior lines of therapy (LOT), had homologous recombination deficiency positive (HRDpos) tumors, had platinum-sensitive disease, and were poly(adenosine 5'-diphosphate [ADP]-ribose) polymerase inhibitors (PARPi) naïve.
Time Frame: Up to 3 years
Population: Primary Analysis Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 47
Percentage of participants | 27.66 [15.6 to 42.6]

2. Secondary Outcome: Duration of Response (DoR)
Description: DoR was defined as the time from first documentation of CR or PR until the time of first documentation of disease progression (PD) as assessed by the Investigator per RECIST (version1.1). DoR was analyzed using Kaplan-Meier (KM) method.
Time Frame: Up to 3 years
Population: Intent-to-Treat (ITT) Population was comprised of all dosed participants with measurable disease at Baseline. Measurable disease at Baseline was determined by the existence of at least 1 target lesion at Baseline tumor scan based on investigator's assessment. Only those participants with data available at the specified time points were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 39
Months | 9.4 [6.6 to 18.3]

3. Secondary Outcome: ORR by HRD Status and Breast Cancer Gene (BRCA) Status
Description: The ORR was defined as the percentage of participants achieving CR or PR as assessed by the Investigator per RECIST (version1.1), where CR=Disappearance of all target lesions. Any pathological lymph nodes must be <10 mm in the short axis. PR=At least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters. ORR was evaluated for participants with following characteristics: HRD status (positive, negative and unknown) and BRCA status (mutation positive, wild-type and unknown).
Time Frame: Up to 3 years
Population: ITT Population. All the participants from the ITT Population were analyzed (461 participants), but only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 461
Percentage of participants
  HRD positive, n=221: number analyzed (Participants) | 221
  HRD positive, n=221 | 14.0 [9.7 to 19.3]
  HRD negative, n=195: number analyzed (Participants) | 195
  HRD negative, n=195 | 2.6 [0.8 to 5.9]
  HRD unknown, n=45: number analyzed (Participants) | 45
  HRD unknown, n=45 | 6.7 [1.4 to 18.3]
  BRCA mutation positive, n=87: number analyzed (Participants) | 87
  BRCA mutation positive, n=87 | 23.0 [14.6 to 33.2]
  BRCA wild-type, n=317: number analyzed (Participants) | 317
  BRCA wild-type, n=317 | 5.0 [2.9 to 8.1]
  BRCA unknown, n=57: number analyzed (Participants) | 57
  BRCA unknown, n=57 | 5.3 [1.1 to 14.6]

4. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease control rate was defined as the percentage of participants achieving CR, PR, or stable disease (SD) as assessed by the Investigator per RECIST (version1.1). The exact (Clopper-Pearson) method was used to calculate 95% confidence interval.
Time Frame: Up to 3 years
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 461
Percentage of participants | 49.02 [44.4 to 53.7]

5. Secondary Outcome: Progression Free Survival
Description: Progression-free survival was defined as the time from the date of first dose to the earlier date of assessment of progression or death by any cause in the absence of progression as assessed by the Investigator per RECIST (version 1.1) or clinical criteria. Progression is defined using RECIST version1.1 as at least a 20% increase in the sum of the diameter of target lesions or unequivocal progression of existing non-target lesions or the appearance of one or more new lesions.
Time Frame: Up to 3 years
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 461
Months | 3.5 [3.2 to 3.7]

6. Secondary Outcome: Overall Survival
Description: Overall Survival was defined as the time from the date of the first dose to the date of death by any cause. It was calculated as (Date of Death minus First dose date plus 1) divided by 30.4375.
Time Frame: Up to 3 years
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 461
Months | 17.2 [14.9 to 19.8]

7. Secondary Outcome: Time to First Subsequent Therapy (TFST)
Description: Time to first subsequent therapy (TFST) was defined as the time from the date of first dose to the date of first subsequent therapy or death, whichever occurs first. It was calculated as (Earlier of [First dose of first subsequent therapy or death] minus First dose date plus 1) divided by 30.4375.
Time Frame: Up to 3 years
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 461
Months | 6.8 [5.9 to 7.5]

8. Other Pre Specified Outcome: Number of Participants With Any Non-serious Adverse Event (Non-SAE) and Any Serious Adverse Event (SAE)
Description: An adverse event is any untoward medical occurrence that occurs in a participant or clinical investigation participant administered a pharmaceutical product, and which does not necessarily have to have a causal relationship with study treatment. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly or birth defect or any other situation according to medical or scientific judgment was categorized as SAE. Adverse events which were not serious were considered as Non-serious adverse events.
Time Frame: Up to a maximum of 71.56 months
Population: Safety Population was comprised of all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 463
Participants
  Any non-SAE | 461
  Any SAE | 200

9. Other Pre Specified Outcome: Number of Participants With Abnormality in Hematology Parameters
Description: Number of participants with abnormality in hematology parameters were planned to be analyzed.
Time Frame: Up to 3 years
Population: Safety Population. This was an other pre-specified outcome measure. Data will not be analyzed and reported.
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: Number of Participants With Abnormality in Clinical Chemistry Parameters
Description: Number of participants with abnormality in clinical chemistry parameters were planned to be analyzed.
Time Frame: Up to 3 years
Population: Safety Population. This was an other pre-specified outcome measure. Data will not be analyzed and reported.
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 0

11. Other Pre Specified Outcome: Number of Participants With Abnormality in Vital Signs
Description: Number of participants with abnormality in vital signs were planned to be analyzed.
Time Frame: Up to 3 years
Population: Safety Population. This was an other pre-specified outcome measure. Data will not be analyzed and reported.
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 0

12. Other Pre Specified Outcome: Number of Participants With Abnormality in Physical Examination
Description: Number of participants with abnormality in physical examination were planned to be analyzed.
Time Frame: Up to 3 years
Population: Safety Population. This was an other pre-specified outcome measure. Data will not be analyzed and reported.
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 0

13. Other Pre Specified Outcome: Number of Participants Who Were Administered Concomitant Medications
Description: Number of participants who were administered concomitant medications were planned to be analyzed.
Time Frame: Up to 3 years
Population: Safety Population. This was an other pre-specified outcome measure. Data will not be analyzed and reported.
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality, Non-serious adverse events (Non-SAEs) and Serious adverse events (SAEs) were reported up to a maximum of 71.56 months
Description: All-cause mortality, Non-SAEs and SAEs were reported for Safety Population which comprised of all participants who received at least 1 dose of study drug.
Arm/Group | Niraparib 300 mg
All-Cause Mortality (participants affected / at risk) | 232/463
Serious Adverse Events (participants affected / at risk) | 200/463
Other Adverse Events (participants affected / at risk) | 461/463
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Niraparib 300 mg (N=463)
Anaemia (Blood and lymphatic system disorders) | 15
Bone marrow failure (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 3
Lymphopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 11
Normochromic anaemia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 34
Arrhythmia supraventricular (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 2
Cardiopulmonary failure (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 2
Pericardial effusion (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Retinal tear (Eye disorders) | 1
Vitreous haemorrhage (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 17
Ascites (Gastrointestinal disorders) | 4
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 10
Diarrhoea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Enteritis (Gastrointestinal disorders) | 1
Erosive oesophagitis (Gastrointestinal disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal fistula (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 2
Intestinal obstruction (Gastrointestinal disorders) | 8
Intestinal perforation (Gastrointestinal disorders) | 1
Large intestinal obstruction (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 21
Obstruction gastric (Gastrointestinal disorders) | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2
Small intestinal obstruction (Gastrointestinal disorders) | 34
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 27
Asthenia (General disorders) | 3
Chest pain (General disorders) | 2
Fatigue (General disorders) | 2
Mucosal inflammation (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 6
Strangulated hernia (General disorders) | 1
Sudden death (General disorders) | 1
Acute hepatic failure (Hepatobiliary disorders) | 1
Biliary tract disorder (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Bacteraemia (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 2
Escherichia urinary tract infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Joint abscess (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Pharyngitis streptococcal (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Pyelonephritis (Infections and infestations) | 2
Sepsis (Infections and infestations) | 8
Streptococcal bacteraemia (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Wound infection (Infections and infestations) | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 2
Electrocardiogram QT prolonged (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 7
Dehydration (Metabolism and nutrition disorders) | 8
Electrolyte imbalance (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 3
Hypophagia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Status epilepticus (Nervous system disorders) | 1
Transient global amnesia (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 2
Nephrolithiasis (Renal and urinary disorders) | 2
Ureteric obstruction (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Deep vein thrombosis (Vascular disorders) | 4
Embolism (Vascular disorders) | 1
Hypertension (Vascular disorders) | 8
Hypotension (Vascular disorders) | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Niraparib 300 mg (N=463)
Anaemia (Blood and lymphatic system disorders) | 233
Anaemia macrocytic (Blood and lymphatic system disorders) | 1
Aplastic anaemia (Blood and lymphatic system disorders) | 1
Increased tendency to bruise (Blood and lymphatic system disorders) | 3
Leukocytosis (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 31
Lymph node pain (Blood and lymphatic system disorders) | 4
Lymphadenopathy (Blood and lymphatic system disorders) | 3
Lymphocytosis (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 15
Neutropenia (Blood and lymphatic system disorders) | 52
Neutrophilia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 151
Thrombocytosis (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 4
Atrial fibrillation (Cardiac disorders) | 5
Atrial flutter (Cardiac disorders) | 1
Atrioventricular block first degree (Cardiac disorders) | 2
Extrasystoles (Cardiac disorders) | 1
Left atrial enlargement (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 34
Pericardial effusion (Cardiac disorders) | 3
Sinus tachycardia (Cardiac disorders) | 14
Tachycardia (Cardiac disorders) | 15
Ventricular arrhythmia (Cardiac disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 3
Auditory disorder (Ear and labyrinth disorders) | 1
Ear congestion (Ear and labyrinth disorders) | 2
Ear discomfort (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 5
Middle ear inflammation (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 3
Vertigo (Ear and labyrinth disorders) | 4
Vestibular disorder (Ear and labyrinth disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Abnormal sensation in eye (Eye disorders) | 1
Age-related macular degeneration (Eye disorders) | 1
Asthenopia (Eye disorders) | 1
Cataract (Eye disorders) | 3
Corneal disorder (Eye disorders) | 1
Diplopia (Eye disorders) | 3
Dry eye (Eye disorders) | 2
Eye disorder (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 2
Night blindness (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Photophobia (Eye disorders) | 2
Photopsia (Eye disorders) | 1
Vision blurred (Eye disorders) | 6
Visual impairment (Eye disorders) | 3
Vitreous floaters (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 10
Abdominal distension (Gastrointestinal disorders) | 68
Abdominal hernia (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 89
Abdominal pain lower (Gastrointestinal disorders) | 11
Abdominal pain upper (Gastrointestinal disorders) | 28
Anal fissure (Gastrointestinal disorders) | 1
Anal haemorrhage (Gastrointestinal disorders) | 1
Anal incontinence (Gastrointestinal disorders) | 1
Anorectal discomfort (Gastrointestinal disorders) | 1
Aphthous ulcer (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 14
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 161
Defaecation urgency (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 81
Dry mouth (Gastrointestinal disorders) | 24
Dyschezia (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 34
Dysphagia (Gastrointestinal disorders) | 7
Epigastric discomfort (Gastrointestinal disorders) | 1
Erosive oesophagitis (Gastrointestinal disorders) | 1
Eructation (Gastrointestinal disorders) | 4
Faeces discoloured (Gastrointestinal disorders) | 2
Faeces hard (Gastrointestinal disorders) | 1
Faeces soft (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 16
Gastric varices (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 26
Gingival bleeding (Gastrointestinal disorders) | 2
Haematemesis (Gastrointestinal disorders) | 2
Haematochezia (Gastrointestinal disorders) | 3
Haemorrhoids (Gastrointestinal disorders) | 5
Hypoaesthesia oral (Gastrointestinal disorders) | 2
Impaired gastric emptying (Gastrointestinal disorders) | 2
Intestinal obstruction (Gastrointestinal disorders) | 3
Large intestinal obstruction (Gastrointestinal disorders) | 4
Lip oedema (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Mouth swelling (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 310
Obstruction gastric (Gastrointestinal disorders) | 1
Odynophagia (Gastrointestinal disorders) | 2
Oesophageal pain (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 4
Oral mucosal erythema (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 3
Paraesthesia oral (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 3
Rectal haemorrhage (Gastrointestinal disorders) | 6
Rectal obstruction (Gastrointestinal disorders) | 1
Rectal spasm (Gastrointestinal disorders) | 1
Retching (Gastrointestinal disorders) | 7
Salivary hypersecretion (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 38
Swollen tongue (Gastrointestinal disorders) | 1
Tongue disorder (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 202
Asthenia (General disorders) | 30
Axillary pain (General disorders) | 1
Chest discomfort (General disorders) | 3
Chest pain (General disorders) | 2
Chills (General disorders) | 13
Drug withdrawal syndrome (General disorders) | 1
Early satiety (General disorders) | 10
Energy increased (General disorders) | 1
Face oedema (General disorders) | 1
Facial pain (General disorders) | 1
Fatigue (General disorders) | 244
Feeling jittery (General disorders) | 2
Gait disturbance (General disorders) | 2
Influenza like illness (General disorders) | 8
Injection site pain (General disorders) | 1
Localised oedema (General disorders) | 2
Malaise (General disorders) | 7
Medical device pain (General disorders) | 1
Mucosal inflammation (General disorders) | 13
Non-cardiac chest pain (General disorders) | 6
Oedema (General disorders) | 3
Oedema peripheral (General disorders) | 31
Pain (General disorders) | 10
Performance status decreased (General disorders) | 1
Peripheral swelling (General disorders) | 15
Pyrexia (General disorders) | 22
Suprapubic pain (General disorders) | 1
Temperature intolerance (General disorders) | 1
Tenderness (General disorders) | 1
Thirst (General disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 2
Drug hypersensitivity (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 2
Seasonal allergy (Immune system disorders) | 8
Abdominal abscess (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Beta haemolytic streptococcal infection (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 8
Candida infection (Infections and infestations) | 3
Cellulitis (Infections and infestations) | 2
Chronic sinusitis (Infections and infestations) | 2
Clostridium difficile infection (Infections and infestations) | 1
Conjunctivitis viral (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Ear infection (Infections and infestations) | 2
Eye infection (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Gingivitis (Infections and infestations) | 1
Hepatitis viral (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 9
Infected cyst (Infections and infestations) | 1
Influenza (Infections and infestations) | 4
Laryngitis (Infections and infestations) | 4
Localised infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 2
Oesophageal candidiasis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 3
Paronychia (Infections and infestations) | 1
Pharyngitis streptococcal (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 7
Pyelonephritis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 2
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 12
Tinea pedis (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 13
Urinary tract infection (Infections and infestations) | 68
Viral infection (Infections and infestations) | 2
Viral upper respiratory tract infection (Infections and infestations) | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 3
Contusion (Injury, poisoning and procedural complications) | 17
Ear canal abrasion (Injury, poisoning and procedural complications) | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 5
Foot fracture (Injury, poisoning and procedural complications) | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Radiation skin injury (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 2
Subarachnoid haemorrhage (Nervous system disorders) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Sunburn (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 17
Alanine aminotransferase increased (Investigations) | 32
Amylase increased (Investigations) | 26
Aspartate aminotransferase increased (Investigations) | 44
Bacterial test positive (Investigations) | 3
Bilirubin conjugated increased (Investigations) | 1
Blood albumin decreased (Investigations) | 7
Blood alkaline phosphatase decreased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 52
Blood bilirubin increased (Investigations) | 10
Blood calcium decreased (Investigations) | 1
Blood chloride decreased (Investigations) | 9
Blood creatine increased (Investigations) | 1
Blood creatinine decreased (Investigations) | 2
Blood creatinine increased (Investigations) | 76
Blood glucose increased (Investigations) | 3
Blood lactate dehydrogenase increased (Investigations) | 15
Blood lactic acid increased (Investigations) | 2
Blood magnesium decreased (Investigations) | 8
Blood potassium decreased (Investigations) | 3
Blood pressure increased (Investigations) | 2
Blood pressure orthostatic decreased (Investigations) | 1
Blood sodium decreased (Investigations) | 4
Blood sodium increased (Investigations) | 1
Blood urea decreased (Investigations) | 1
Blood urea increased (Investigations) | 11
Blood urine present (Investigations) | 3
Carbohydrate antigen 125 increased (Investigations) | 1
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 21
Gamma-glutamyltransferase increased (Investigations) | 50
Glomerular filtration rate abnormal (Investigations) | 1
Glomerular filtration rate decreased (Investigations) | 4
Glomerular filtration rate increased (Investigations) | 1
Glucose tolerance test abnormal (Investigations) | 1
Glucose urine present (Investigations) | 1
Haemoglobin decreased (Investigations) | 6
Haemoglobin urine present (Investigations) | 4
Heart rate increased (Investigations) | 3
International normalised ratio increased (Investigations) | 6
Lymphocyte count decreased (Investigations) | 32
Lymphocyte count increased (Investigations) | 1
Mean cell volume increased (Investigations) | 2
Mean platelet volume decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 39
Neutrophil count increased (Investigations) | 2
Nitrite urine present (Investigations) | 2
Platelet count decreased (Investigations) | 101
Platelet count increased (Investigations) | 2
Protein total decreased (Investigations) | 6
Protein total increased (Investigations) | 2
Protein urine present (Investigations) | 10
Prothrombin time prolonged (Investigations) | 6
QRS axis abnormal (Investigations) | 2
Urine ketone body present (Investigations) | 2
Urine leukocyte esterase (Investigations) | 3
Urine leukocyte esterase positive (Investigations) | 8
Vitamin D decreased (Investigations) | 1
Weight decreased (Investigations) | 45
Weight increased (Investigations) | 2
White blood cell count decreased (Investigations) | 56
White blood cell count increased (Investigations) | 2
White blood cells urine positive (Investigations) | 4
Appetite disorder (Metabolism and nutrition disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 127
Dehydration (Metabolism and nutrition disorders) | 44
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 34
Hyperkalaemia (Metabolism and nutrition disorders) | 10
Hypermagnesaemia (Metabolism and nutrition disorders) | 3
Hypernatraemia (Metabolism and nutrition disorders) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Hypervolaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 25
Hypocalcaemia (Metabolism and nutrition disorders) | 17
Hypochloraemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 39
Hypomagnesaemia (Metabolism and nutrition disorders) | 91
Hyponatraemia (Metabolism and nutrition disorders) | 52
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Hypoproteinaemia (Metabolism and nutrition disorders) | 1
Iron deficiency (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 24
Back pain (Musculoskeletal and connective tissue disorders) | 50
Costochondritis (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 9
Groin pain (Musculoskeletal and connective tissue disorders) | 6
Joint swelling (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 16
Muscle twitching (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 19
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 11
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 17
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 17
Neck pain (Musculoskeletal and connective tissue disorders) | 9
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18
Pain in jaw (Musculoskeletal and connective tissue disorders) | 3
Spondylitis (Musculoskeletal and connective tissue disorders) | 1
Trismus (Musculoskeletal and connective tissue disorders) | 2
Metastases to breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Akathisia (Nervous system disorders) | 1
Amnesia (Nervous system disorders) | 1
Anosmia (Nervous system disorders) | 3
Aphasia (Nervous system disorders) | 1
Ataxia (Nervous system disorders) | 1
Balance disorder (Nervous system disorders) | 3
Cognitive disorder (Nervous system disorders) | 2
Coordination abnormal (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 52
Dizziness postural (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 19
Extrapyramidal disorder (Nervous system disorders) | 1
Headache (Nervous system disorders) | 89
Hypoaesthesia (Nervous system disorders) | 7
Hypogeusia (Nervous system disorders) | 1
Hyposmia (Nervous system disorders) | 2
Lethargy (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Loss of proprioception (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 5
Migraine (Nervous system disorders) | 1
Monoplegia (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 14
Paraesthesia (Nervous system disorders) | 4
Parosmia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 10
Post-traumatic headache (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Restless legs syndrome (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 4
Secondary cerebellar degeneration (Nervous system disorders) | 1
Sinus headache (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 4
Tremor (Nervous system disorders) | 6
Vocal cord paralysis (Nervous system disorders) | 1
Device occlusion (Product Issues) | 2
Abnormal dreams (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 38
Confusional state (Psychiatric disorders) | 11
Depression (Psychiatric disorders) | 17
Insomnia (Psychiatric disorders) | 105
Mania (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 2
Nervousness (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 3
Bladder discomfort (Renal and urinary disorders) | 2
Bladder spasm (Renal and urinary disorders) | 1
Chromaturia (Renal and urinary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 6
Dysuria (Renal and urinary disorders) | 10
Glycosuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 12
Hydronephrosis (Renal and urinary disorders) | 6
Incontinence (Renal and urinary disorders) | 3
Micturition urgency (Renal and urinary disorders) | 6
Pollakiuria (Renal and urinary disorders) | 9
Proteinuria (Renal and urinary disorders) | 15
Renal failure (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Renal pain (Renal and urinary disorders) | 1
Ureteric obstruction (Renal and urinary disorders) | 1
Urethral pain (Renal and urinary disorders) | 2
Urinary hesitation (Renal and urinary disorders) | 2
Urinary incontinence (Renal and urinary disorders) | 5
Urinary retention (Renal and urinary disorders) | 2
Urinary tract pain (Renal and urinary disorders) | 3
Urine abnormality (Renal and urinary disorders) | 1
Urine odour abnormal (Renal and urinary disorders) | 2
Urogenital disorder (Renal and urinary disorders) | 1
Adnexa uteri pain (Reproductive system and breast disorders) | 1
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1
Breast disorder (Reproductive system and breast disorders) | 1
Breast mass (Reproductive system and breast disorders) | 1
Breast pain (Reproductive system and breast disorders) | 3
Breast swelling (Reproductive system and breast disorders) | 1
Cystocele (Reproductive system and breast disorders) | 1
Nipple pain (Reproductive system and breast disorders) | 1
Pelvic discomfort (Reproductive system and breast disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 4
Vaginal discharge (Reproductive system and breast disorders) | 6
Vaginal disorder (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 6
Vulvovaginal discomfort (Reproductive system and breast disorders) | 2
Vulvovaginal dryness (Reproductive system and breast disorders) | 1
Vulvovaginal erythema (Reproductive system and breast disorders) | 1
Vulvovaginal pain (Reproductive system and breast disorders) | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 64
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 88
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 23
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 22
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 18
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3
Acne cystic (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 18
Blood blister (Skin and subcutaneous tissue disorders) | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 7
Ecchymosis (Skin and subcutaneous tissue disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6
Madarosis (Skin and subcutaneous tissue disorders) | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 8
Onychoclasis (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 8
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 9
Purpura (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 19
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Skin mass (Skin and subcutaneous tissue disorders) | 1
Skin tightness (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2
Tooth extraction (Surgical and medical procedures) | 1
Angiopathy (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 3
Embolism (Vascular disorders) | 4
Flushing (Vascular disorders) | 5
Haematoma (Vascular disorders) | 2
Hot flush (Vascular disorders) | 21
Hypertension (Vascular disorders) | 60
Hypotension (Vascular disorders) | 5
Lymphoedema (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Peripheral coldness (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 2
Venous occlusion (Vascular disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Bundle branch block right (Cardiac disorders) | 2
Coronary artery disease (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 3
Paraesthesia ear (Ear and labyrinth disorders) | 1
Hyperparathyroidism (Endocrine disorders) | 1
Eye pruritus (Eye disorders) | 1
Scleral discolouration (Eye disorders) | 1
Abdominal rigidity (Gastrointestinal disorders) | 1
Gastric mucosa erythema (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Oesophageal stenosis (Gastrointestinal disorders) | 1
Complication associated with device (General disorders) | 1
Cyst (General disorders) | 1
Swelling (General disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
COVID-19 (Infections and infestations) | 1
Helicobacter infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 16
Otitis externa (Infections and infestations) | 1
Perineal abscess (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Vulval abscess (Infections and infestations) | 2
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Blood cholesterol increased (Investigations) | 1
Lipase increased (Investigations) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ageusia (Nervous system disorders) | 1
Dyskinesia (Nervous system disorders) | 1
Head titubation (Nervous system disorders) | 1
Taste disorder (Nervous system disorders) | 3
Panic attack (Psychiatric disorders) | 1
Ureterolithiasis (Renal and urinary disorders) | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT02354586/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT02354586/SAP_002.pdf